CLINICAL TRIAL: NCT05761847
Title: Optimizing the Clinical Management of Polypharmacy for Children With Medical Complexity: The Pediatric Medication Therapy Management (pMTM) Trial
Brief Title: Pediatric Medication Therapy Management Trial
Acronym: pMTM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-2423; 1R01HS028979-01A1 (AHRQ)
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Child, Only; Disabilities Multiple; Medication Interaction; Medication Compliance; Medication Administered in Error
Keywords: Children with Medical Complexity; Polypharmacy; Medication Safety
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Hybrid Type 2 Randomized Controlled Trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The usual care group will receive standard-of-care medication management practices delivered during the course of a routine clinical visit.
- Intervention (Experimental): The intervention group will receive the pMTM study intervention before a routine clinical visit.
  Interventions: Other: Pediatric Medication Therapy Management (pMTM)

INTERVENTIONS:
Other: Pediatric Medication Therapy Management (pMTM) — The pMTM intervention is comprised of 3 activities: comprehensive review of the medication regimen; optimization of the medication regimen; and creation of the medication action plan.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate whether an intervention called Pediatric Medication Therapy Management (pMTM) improves the identification and management of medication-related problems among children with medical complexity and polypharmacy.

DETAILED DESCRIPTION:
Patients and their parents who meet the study eligibility requirements will be invited to participate in the study. After being informed about the study and potential risks, all patients and their parents giving written informed consent (and assent, when appropriate) will be randomized in a 1:1 ratio to usual care or to the Pediatric Medication Therapy Management (pMTM) intervention.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* ≥1 complex chronic condition (CCC)
* ≥5 current medications (including prescription, as needed, and over-the-counter medications)
* Receives primary care at Children's Hospital Colorado

Exclusion Criteria:

* Non-English speaking
* Sibling or family member already enrolled in this study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 371 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Medication-Related Problem (MRP) Count | 90 Days
  A MRP is a clearly defined event involving medication therapy that interferes with an optimum outcome for a specific patient, including: inappropriate or unnecessary therapy; suboptimal therapy; undertreated symptom; adverse drug event; major drug-drug interaction; duplication of therapy; or, unclear prescription instruction.

SECONDARY OUTCOMES:
Change in Parent-Reported Outcomes of Symptoms (PRO-Sx) Global Symptom Score | Baseline and 90 Days
  The PRO-Sx instrument assesses 28 physical and psychological symptoms over the past week. The study instrument is designed to be completed by a full-proxy parent and contains 28 symptom items, each with 4-point scores for domains of frequency, severity, and extent of bother. Based on these components, a global symptom score and individual symptom scores can be calculated (0-100 scale, with 100 being the worst). Change equals the 90-day score minus the baseline score.
Acute Healthcare Visit Count | 90 Days
  Unplanned acute healthcare visits include: ambulatory sick visits; emergency room visits; and, inpatient hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: James A Feinstein, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feinstein JA, Friedman H, Orth LE, Feudtner C, Kempe A, Samay S, Blackmer AB. Complexity of Medication Regimens for Children With Neurological Impairment. JAMA Netw Open. 2021 Aug 2;4(8):e2122818. doi: 10.1001/jamanetworkopen.2021.22818. PMID 34436607
- [Background] Marquez C, Thompson R, Feinstein JA, Orth LE. Identifying opportunities for pediatric medication therapy management in children with medical complexity. J Am Pharm Assoc (2003). 2022 Sep-Oct;62(5):1587-1595.e3. doi: 10.1016/j.japh.2022.04.005. Epub 2022 Apr 12. PMID 35527209
- [Background] Feinstein JA, Hall M, Antoon JW, Thomson J, Flores JC, Goodman DM, Cohen E, Azuine R, Agrawal R, Houtrow AJ, DeCourcey DD, Kuo DZ, Coller R, Gaur DS, Berry JG. Chronic Medication Use in Children Insured by Medicaid: A Multistate Retrospective Cohort Study. Pediatrics. 2019 Apr;143(4):e20183397. doi: 10.1542/peds.2018-3397. PMID 30914443
- [Background] Feinstein JA, Feudtner C, Blackmer AB, Valuck RJ, Fairclough DL, Holstein J, Gregoire L, Samay S, Kempe A. Parent-Reported Symptoms and Medications Used Among Children With Severe Neurological Impairment. JAMA Netw Open. 2020 Dec 1;3(12):e2029082. doi: 10.1001/jamanetworkopen.2020.29082. PMID 33306117
- [Background] Feinstein JA, Feudtner C, Valuck RJ, Fairclough DL, Holstein JA, Samay S, Kempe A. Identifying Important Clinical Symptoms in Children With Severe Neurological Impairment Using Parent-Reported Outcomes of Symptoms. JAMA Pediatr. 2020 Nov 1;174(11):1114-1117. doi: 10.1001/jamapediatrics.2020.2987. PMID 33044500
- [Result] Orth LE, Feudtner C, Kempe A, Morris MA, Colborn KL, Gritz RM, Linnebur SA, Begum A, Feinstein JA. A coordinated approach for managing polypharmacy among children with medical complexity: rationale and design of the Pediatric Medication Therapy Management (pMTM) randomized controlled trial. BMC Health Serv Res. 2023 Apr 29;23(1):414. doi: 10.1186/s12913-023-09439-y. PMID 37120509

DOCUMENTS (1):
  • Informed Consent Form (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT05761847/ICF_000.pdf